CLINICAL TRIAL: NCT02530879
Title: Comparison of Voice Therapy and Antireflex Therapy in the Treatment of Laryngopharyngeal Reflux-related Hoarseness: A Prospective Randomized Control Trial
Brief Title: Comparison of Voice Therapy and Antireflex Therapy in LPR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 22455
Record Dates: First submitted 2015-08-06; First posted 2015-08-21 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Omeprazole; Lansoprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voice therapy (Experimental): Evaluation is completed over two, one-hour sessions. Once the evaluation is complete, the subject will begin weekly, individual voice therapy for 55 minute sessions per week with a second year graduate student under the direct supervision of the clinical faculty member.Treatment sessions will include a counseling component and an active exercise program.
  Interventions: Behavioral: Voice therapy
- Antireflux medication (Active Comparator): Intervention includes treatment with one of the following:
  1. Omeprazole- Dose range oral, 20mg once a day, up to 40mg twice a day
  2. Lansoprazole-Dose range 15mg per day- 30mg twice a day
  3. Esomeprazole- Dose range oral, 20mg once a day, up to 40mg twice a day
  4. Rantidine-Dose range: 150 mg twice a day or 300 mg once a day.
  5. Rantidine may be used in combination with any of the above
  Interventions: Drug: Omeprazole, Lansoprazole, Esomeprazole, Rantidine
- Voice therapy and Anti-reflux therapy (Experimental): Subjects will receive both anti-reflux medication as detailed above and voice therapy as detailed above.
  Interventions: Other: Combination of anti-reflux medication and voice therapy

INTERVENTIONS:
Drug: Omeprazole, Lansoprazole, Esomeprazole, Rantidine — 1.Omeprazole- Dose range oral, 20mg once a day, up to 40mg twice a day 2.Lansoprazole-Dose range 15mg per day- 30mg twice a day 3.Esomeprazole- Dose range oral, 20mg once a day, up to 40mg twice a day 4.Rantidine-Dose range: 150 mg twice a day or 300 mg
  Arms: Antireflux medication
Behavioral: Voice therapy — Evaluation is completed over two, one-hour sessions. Once the evaluation is complete, the subject will begin weekly, individual voice therapy for 55 minute sessions per week with a second year graduate student under the direct supervision of the clinical faculty member.Treatment sessions will include a counseling component and an active exercise program.
  Arms: Voice therapy
Other: Combination of anti-reflux medication and voice therapy — Subjects will receive both anti-reflux medication as detailed above and voice therapy as detailed above.
  Arms: Voice therapy and Anti-reflux therapy

SUMMARY:
This study will be a prospective, randomized, unblinded but controlled trial. Patients presenting to the Otolaryngology clinic who are diagnosed with laryngopharyngeal reflux disorder related dysphonia and meet inclusion criteria will be eligible to enroll in the study. Subjects will be randomized to one of three treatment arms, voice therapy, anti-reflux therapy, or a combination of voice therapy and anti-reflux therapy. Reflux symptom index (RSI) scores, reflux finding scores (RFS), voice handicap index-10 (VHI-10) scores, and consensus auditory perceptual evaluation-voice (CAPE-V) scores will be compared prior to initiation of therapy as well as at 1, 2, and 3 months following initiation of treatment.

DETAILED DESCRIPTION:
Hoarseness is one of the most common presenting complaints in otolaryngology. The differential diagnosis for hoarseness is board, but a large percentage has been attributed to laryngopharyngeal reflux (LPR). LPR refers to the symptomatic effects of regurgitated gastric contents into the pharynx and larynx.1-3 1,2 Although dual-probe 24 hour pH monitoring is the gold standard in the diagnosis of LPR, it is not always performed due to inconvenience and cost. Patients are commonly treated based on history and physical examination findings alone. The literature on the efficacy of anti-reflux therapy and LPR is controversial. Karkos et al performed a systematic review on the use of empiric treatment of proton pump inhibitors (PPI) in patients suspected of having LPR and found no statistically significant difference between patients treated with PPI and those treated with placebo in reference to symptom severity or frequency of presumed reflux events. 2 Commonly patients are started on empiric therapy with anti-reflux medications and lifestyle modifications. Laryngoscopy is performed on all patients presenting with dysphonia. While a variety of findings have been characterized as consistent with reflux a study performed by Hicks et al, found that 86% of normal volunteers had findings consistent with reflux on flexible laryngoscopy.5 This calls into question the sensitivity and specificity of laryngoscopy in the diagnosis of LPR. Park et al performed a study comparing the effectiveness of anti-reflux therapy alone versus a combination of voice therapy with PPI in the treatment of presumed LPR-related dysphonia, and found combination therapy to be superior to anti-reflux therapy alone. 3 Because there are no studies comparing voice therapy directly with anti-reflux therapy, one cannot determine whether the improvements are due to augmentation of anti-reflux therapy with voice therapy, or if voice therapy alone is superior in the treatment of LPR-related dysphonia. There are currently no studies comparing the effectiveness of voice therapy alone, anti-reflux therapy alone, and combination therapy. Patients who present with dysphonia may be over treated with anti-reflux medications. These medications are not without side effects. It is hypothesized that a subset of patients who are thought to have reflux related dysphonia are misusing their voice and can be successfully treated with voice therapy alone. This study will be a prospective, randomized, unblinded but controlled trial. Patients presenting to the Otolaryngology clinic who are diagnosed with LPR-related dysphonia who meet inclusion criteria will be eligible to enroll in the study and will be randomized to one of the three treatment arms. Reflux symptom index (RSI) scores, reflux finding scores (RFS), voice handicap index-10 (VHI-10) scores, and consensus auditory perceptual evaluation-voice (CAPE-V) scores will be compared prior to initiation of therapy as well as at 1, 2, and 3 months following initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Hoarseness
* Reflux symptom index score >13
* Reflux finding score >7
* English speaking

Exclusion Criteria:

* Evidence of other laryngeal pathology
* Esophageal dysmotility
* Gastroesophageal reflux
* Currently on anti-reflux medications
* Presence of a neurologic condition
* Active smoking
* Currently pregnant
* Individuals unable to consent for themselves
* Recent upper respiratory infection lasting more than 1 month
* Prior treatment for laryngopharyngeal reflux.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of pre and post treatment voice outcomes in LPR-related dysphonia based on pre and post treatment CAPE-V Scores | 3 months
  Voice outcomes in patients with LPR related dysphonia treated with voice therapy, anti-reflux therapy, or a combination will be compared based on consensus auditory perceptual evaluation-voice scores
Comparison of treatment outcomes in laryngeal reflux findings based on RFS scores | 3 months
  Reflux finding scores based on laryngoscopy findings will be obtained at the beginning of the study and after treatment. Subjects treated with voice therapy, anti-reflux medication, or a combination will be compared.
Comparison of treatment outcomes in laryngeal reflux symptoms based on RSI scores | 3 months
  Reflux symptom index is a questionnaire subjects will fill out before the study and after treatment. Subjects treated with voice therapy, anti-reflux medication, or a combination will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nausheen Jamal, MD, Principal Investigator — Temple Hospital faculty member
Locations (2):
- United States (2):
  - Temple Otolaryngology, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with participants at the completion of the 3 month study period

REFERENCES:
- [Background] Fusconi M, De Virgilio A, Conte M, Colicchio MG, Gallo A, Greco A, Ralli G, de Vincentiis M. The importance of the number of reflux episodes in the diagnosis of laryngopharyngeal reflux disease. Otolaryngol Head Neck Surg. 2013 Feb;148(2):261-6. doi: 10.1177/0194599812466534. Epub 2012 Nov 2. PMID 23124925
- [Background] Hicks DM, Ours TM, Abelson TI, Vaezi MF, Richter JE. The prevalence of hypopharynx findings associated with gastroesophageal reflux in normal volunteers. J Voice. 2002 Dec;16(4):564-79. doi: 10.1016/s0892-1997(02)00132-7. PMID 12512644
- [Result] Koufman JA, Aviv JE, Casiano RR, Shaw GY. Laryngopharyngeal reflux: position statement of the committee on speech, voice, and swallowing disorders of the American Academy of Otolaryngology-Head and Neck Surgery. Otolaryngol Head Neck Surg. 2002 Jul;127(1):32-5. doi: 10.1067/mhn.2002.125760. No abstract available. PMID 12161727
- [Result] Karkos PD, Wilson JA. Empiric treatment of laryngopharyngeal reflux with proton pump inhibitors: a systematic review. Laryngoscope. 2006 Jan;116(1):144-8. doi: 10.1097/01.mlg.0000191463.67692.36. PMID 16481828
- [Result] Park JO, Shim MR, Hwang YS, Cho KJ, Joo YH, Cho JH, Nam IC, Kim MS, Sun DI. Combination of voice therapy and antireflux therapy rapidly recovers voice-related symptoms in laryngopharyngeal reflux patients. Otolaryngol Head Neck Surg. 2012 Jan;146(1):92-7. doi: 10.1177/0194599811422014. Epub 2011 Sep 9. PMID 21908799